CLINICAL TRIAL: NCT04861376
Title: Pueraria Lobata and Pueraria Thomsonii for Mild Dyslipidemia: A Double-blinded Randomized Placebo-controlled Trial
Brief Title: Pueraria Lobata and Pueraria Thomsonii for Mild Dyslipidemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangxi University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Xu Zhou, Associated professor, Jiangxi University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JXUTCM-EBM-04
Record Dates: First submitted 2021-04-24; First posted 2021-04-27 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Dyslipidemias
Keywords: Dyslipidemias, Pueraria lobata, Pueraria thomsonii
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pueraria lobata group (Experimental): Pueraria lobata will be made into granules.
  Interventions: Drug: Pueraria lobata
- Pueraria thomsoni group (Experimental): Pueraria thomsoni will be made into granules.
  Interventions: Drug: Pueraria thomsoni
- Placebo group (Placebo Comparator): The dosage form, specifications and packaging of the placebo will be no different from those of Pueraria lobata and Pueraria thomsoni Granules, and the smell and taste will be basically the same.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pueraria lobata — The dose of Pueraria lobata granules is one sachet per day, 1.5g per sachet, which equivalent to 15g of the original drug.
  Arms: Pueraria lobata group
Drug: Pueraria thomsoni — The dose of Pueraria thomsoni granules is one sachet per day, 1.5g per sachet, which equivalent to 15g of the original drug.
  Arms: Pueraria thomsoni group
Other: Placebo — The placebo group will take the same dose as the other two groups.
  Arms: Placebo group

SUMMARY:
Dyslipidemia is an important risk factor for atherosclerotic cardiovascular disease. Maintaining normal levels of lipid indicators can significantly reduce the risk of atherosclerotic cardiovascular disease and mortality. Empirical evidence suggests that adherence to Pueraria lobata and Pueraria thomsonii is useful for improving dyslipidemia, but evidence from randomized controlled trials is lacking. This randomized, double-blind controlled trial is therefore designed to evaluate the efficacy and safety of Pueraria lobata and Pueraria thomsonii for dyslipidemia.

DETAILED DESCRIPTION:
Pueraria is an important Chinese herbal medicine. The Pharmacopoeia of the People's Republic of China classifies the Pueraria as Pueraria lobata and Pueraria thomsonii according to the different sources of the plant, both of them is sweet, pungent and cool in nature, and has the effects of relieving fever, quenching thirst, penetrating rashes, raising the Yang to stop diarrhea, activating the meridians and detoxifying alcohol. As early as in the Han Dynasty, Zhongjing Zhang's "Treatise on Febrile Diseases" described the famous formula "Pueraria Tang", which is still an important formula for relieving exterior syndromes.

In clinical practice, the preparations of Pueraria lobata and Pueraria thomsonii are widely used to treat headache, dizziness, hypertension, coronary heart disease, angina pectoris, myocardial infarction and other diseases. For example, the puerarin injection has the effects of dilating blood vessels, slowing down heart rate, reducing myocardial oxygen consumption and improving blood circulation in the heart and brain.

Although the puerarin has been shown to be effective in a variety of cardiovascular diseases, as of now, it is unclear whether Pueraria lobata and Pueraria thomsonii can be used as part of the daily diet to regulate blood lipids and improve dyslipidemia. Therefore, the aim of this study is to conduct a randomized, double-blind controlled trial that includes patients with mildly elevated lipids to evaluate the efficacy and safety of Pueraria lobata and Pueraria thomsonii for dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Marginally elevated low-density lipoprotein (LDL-C), 3.4 to 4.1 mmol/L
* Informed consent to the study and signed the informed consent form

Exclusion Criteria:

* Patients who have a history of allergy to Pueraria Lobata or Pueraria Thomsonii.
* Patients who have taken lipid-lowering drugs within a week
* Patients with secondary dyslipidemia caused by other diseases or medications taken.
* Pregnant or lactating women.
* Patients who combine cognitive dysfunction, disorders of consciousness, psychiatric disorders, dyslexia or verbal communication dysfunction
* Patients with a combination of other serious diseases, such as malignant tumors, hepatic or renal insufficiency, cardiovascular or cerebrovascular disease, etc.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2021-06-05 (Actual); Primary Completion 2022-01-22 (Actual); Study Completion 2022-01-22 (Actual)

PRIMARY OUTCOMES:
Low-density lipoprotein cholesterol | Baseline, month 1, and month 3
  Change from baseline in low-density lipoprotein cholesterol level

SECONDARY OUTCOMES:
High-density lipoprotein cholesterol | Baseline, month 1, and month 3
  Change from baseline in high-density lipoprotein cholesterol level
Triglyceride | Baseline, month 1, and month 3
  Change from baseline in triglyceride level
Total cholesterol | Baseline, month 1, and month 3
  Change from baseline in total cholesterol level
Systolic blood pressure | Baseline, month 1, and month 3
  Changes in systolic blood pressure
Diastolic blood pressure | Baseline, month 1, and month 3
  Changes in diastolic blood pressure
Fasting blood glucose | Baseline, month 1, and month 3
  Changes in fasting blood glucose
Symptoms related to dyslipidemia | Baseline, month 1, and month 3
  Symptoms related to dyslipidemia that is measured by a Standardized Chinese Medicine Physical Fitness Scale
Serum metabolomics | Baseline, month 1, and month 3
  To identify changes in in plasma (or serum) endogenous components between patients with dyslipidemia, find biomarkers, and explore the modulation of various biomarkers after taking Pueraria Lobata and Pueraria Thomsonii
Urine metabolomics | Baseline, month 1, and month 3
  To identify changes in urine endogenous components between patients with dyslipidemia, find biomarkers, and explore the modulation of various biomarkers after taking Pueraria Lobata and Pueraria Thomsonii
Any adverse events | Baseline, month 1, and month 3
  An adverse event is defined as any medically induced harm, including preventable and nonpreventable adverse events. In this study, adverse events also included those in which blood, urine, stool routine, cardiac, liver and kidney function, and the four coagulation tests exceeded or fell below two times normal values or judged by the physician to be clinically significant abnormal values.
Any severe adverse events | Baseline, month 1, and month 3
  Severe adverse events refer to events requiring hospitalization, prolonged hospitalization, disability, impact on work capacity, life-threatening or death that occur during clinical trials.
Treatment-related adverse events | Baseline, month 1, and month 3
  The relationship will be judged based on a combination of the following criteria: 1) there is a logical sequence in time and space between the adverse reaction and the mydriatic intervention; 2) the adverse reaction cannot be explained by other combined treatments or comorbidities; the symptoms of the adverse reaction resolved or disappeared after discontinuation of the intervention; 3) the causal association between the adverse reaction and the intervention is supported by an established pharmacological or phenomenological mechanism; and 4) the reappearance of the adverse event is triggered by reapplication of the drug.
Withdrawal due to adverse events | Baseline, month 1, and month 3
  Withdrawal due to any adverse events will be counted.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Nanchang Hongdu Hospital of Traditional Chinese Medicine, Nanchang, Jiangxi
  - The Affiliated Hospital of Jiangxi University of Chinese Medicine, Nanchang, Jiangxi

IPD SHARING:
Plan to Share IPD: No